CLINICAL TRIAL: NCT06148272
Title: A Single-ascending and Multiple-ascending Dose Study of LY3971297 in Healthy Participants and Participants With Obesity and Hypertension and Participants With Decreased Estimated Glomerular Filtration Rate
Brief Title: A Study of LY3971297 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18771; J4O-MC-EZHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY3971297 (Part A) (Experimental): Single ascending doses of LY3971297 administered subcutaneously (SC) in healthy participants
  Interventions: Drug: LY3971297
- LY3971297 (Part B) (Experimental): Multiple ascending doses of LY3971297 administered SC in healthy participants
  Interventions: Drug: LY3971297
- LY3971297 (Part C) (Experimental): Multiple ascending doses of LY3971297 administered SC in healthy Chinese participants
  Interventions: Drug: LY3971297
- LY3971297 (Part D) (Experimental): Multiple ascending doses of LY3971297 administered SC
  Interventions: Drug: LY3971297
- LY3971297 (Part E) (Experimental): Multiple doses of LY3971297 administered SC in healthy Japanese participants
  Interventions: Drug: LY3971297
- Placebo (Part A, B, C, D, E, & G) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3971297 (Part F) (Experimental): Single doses of LY3971297 administered intravenously (IV) in healthy participants
  Interventions: Drug: LY3971297 IV
- LY3971297 (Part G) (Experimental): Multiple doses of LY3971297 administered SC
  Interventions: Drug: LY3971297

INTERVENTIONS:
Drug: LY3971297 — Administered SC
  Arms: LY3971297 (Part A); LY3971297 (Part B); LY3971297 (Part C); LY3971297 (Part D); LY3971297 (Part E); LY3971297 (Part G)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A, B, C, D, E, & G)
Drug: LY3971297 IV — Administered IV
  Arms: LY3971297 (Part F)

SUMMARY:
The purpose of this study is to measure side effects of LY3971297 injection administered under the skin in healthy participants and obese participants with high blood pressure (BP). Blood tests will be performed to check how much LY3971297 gets into the bloodstream and how long it takes the body to eliminate it. This is a 7-part study. The study duration will be approximately 60 days for Parts A and F, and approximately 90 days for Parts B, C, D, E, and G.

ELIGIBILITY:
Inclusion Criteria:

* For Parts A, B, C, E, and F: Overtly healthy males or females as determined by medical history and physical examination
* For Parts A, B, C, E, and F: Have a screening body mass index (BMI) in the range of 18.5 to 35 kilogram per square meter (kg/m²), inclusive, with no significant weight gain or loss in the past 3 months prior to screening
* For Part C, to qualify as Chinese for the purpose of this study, all the participants' biological grandparents must be of exclusive Chinese descent and born in China
* For Part D, participants must have a stable dose of medications within the past 3 months prior to screening
* For Part D, obesity BMI in the range of 30 to 40 kg/m², inclusive, with a waist circumference of at least 102 centimeter (cm) for men and at least 89 cm for women for participants of US sites only. For participants of Singaporean, South Asian, Japanese, and/or Chinese Origin at sites outside the US, the BMI range is 27 to 40 kg/m2 and the waist circumference is at least 90 cm for men and at least 80 cm for women
* For Part E, to qualify as a participant of the first-generation Japanese origin, the participant, the participant's biological parents, and all of the participants' biological grandparents must be of exclusive Japanese descent and born in Japan
* Male participants must agree to adhere to contraception restrictions and female participants must be women not of childbearing potential
* For Part G, have a screening BMI in the range of 18.5 to 40 kg/m², inclusive, with no significant weight gain or loss in the past 3 months prior to screening
* For Part G, participants have a decreased estimated glomerular filtration rate (eGFR)
* For Parts D and G, participants are allowed to have stable background treatment for hypertension, type 2 diabetes mellitus (on oral drug therapy and/or long-acting insulin), dyslipidemia (on statin therapy) and/or hypothyroidism as determined by the investigator
* For Part G, Participants should be on a stable dose of angiotensin converting enzyme inhibitor or angiotensin II receptor blocker

Exclusion Criteria:

* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Have known or ongoing psychiatric disorders that, in the opinion of the investigator, increases the risks associated with study participation
* Have blood pressure and/or pulse rate constituting a risk as determined by the investigator
* Have a systolic blood pressure (BP) of less than 100 millimeters of mercury (mmHg)
* Diagnosed with orthostatic hypotension defined as a decrease in systolic blood pressure of equal to or greater than 20 mmHg or a decrease in diastolic blood pressure of equal to or greater than 10 mmHg when compared with BP from the supine position
* For US sites: have donated blood of more than 500 mL within the previous 3 months of screening or intend to donate blood during the course of the study
* For Singapore sites: Have donated blood of more than 450 mL or more in the past 3 months or provided any blood donation within the past 1 month before screening
* Consume more than 10 cigarettes per day (or the equivalent) or are unable or unwilling to abstain from nicotine
* Have alcohol intake that exceeds recommended alcohol consumption limits per local regulation or are unwilling to stop alcohol consumption 24 hours prior to dosing until discharge
* For Part D, has concurrent use or anticipated use of phosphodiesterase 5 inhibitor such as vardenafil, tadalafil, and sildenafil, soluble guanylyl cyclase activators (such as riociguat and vericiguat)
* For Parts D and G, has concurrent or anticipated use of long-acting nitrates or nitric oxide (NO) donors
* For Part D, has current use of more than 3 mechanism of actions for treatment of hypertension
* For Part G, has previous or current diagnosis of primary glomerulopathy, vasculitic renal disease, prior dialysis or unstable rapidly progressing renal disease, autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis, or anti-neutrophil cytoplasm antibody-associated vasculitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Part A and F: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline (Day of Exposure) to Day 29 post-dose
  Part A and F: A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module
Part B, C, D, E, & G: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline (Day of Exposure) to Day 57 post-dose
  Part B, C, D, E, & G: A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module
Part F: Pharmacokinetics (PK): Area Under the Concentration curve (AUC) of LY3971297 | Baseline Up to Day 29 post-dose for Part F
  Part F: PK: AUC of LY3971297
Part F: PK: Maximum Observed Drug Concentration (Cmax) of LY3971297 | Baseline Up to Day 29 post-dose for Part F
  Part F: PK: Cmax of LY3971297

SECONDARY OUTCOMES:
Part B, C, D, E, and G: Pharmacokinetics (PK): Area Under the Concentration curve (AUC) of LY3971297 | Predose on day 1 up to 29 days post-dose for Part A and pre-dose on day 1 up to 57 days post-dose for Part B, C, D, E, and G
  Part B, C, D, E, and G: PK: AUC of LY3971297
Part B, C, D, E, and G: PK: Maximum Observed Drug Concentration (Cmax) of LY3971297 | Predose on day 1 up to 29 days post-dose for Part A and pre-dose on day 1 up to 57 days post-dose for Part B, C, D, E, and G
  Part B, C, D, E, and G: PK: Cmax of LY3971297

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (2):
  - CenExel ACT, Anaheim, California
  - ICON Early Phase Services, San Antonio, Texas
- Japan (3):
  - Hakata Clinic, Fukuoka
  - P-One Clinic, Hachiōji
  - Clinical Research Hospital Tokyo, Shinjuku-ku
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No